CLINICAL TRIAL: NCT05251480
Title: Examining the Effectiveness of DermGEN™ Versus Standard of Care in the Treatment of Diabetic Foot Ulcers in First Nations People Living in Northwestern Ontario Communities
Brief Title: Examining the Effectiveness of DermGEN™ in the Treatment of Diabetic Foot Ulcers in First Nations People
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DeCell Technologies Inc. (Industry)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Dalhousie University (Other); Lakehead University (Other)
Responsible Party: Principal Investigator, Dr. Paul F. Gratzer, Associate Professor, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DermGEN.RCT-01
Record Dates: First submitted 2021-11-03; First posted 2022-02-22 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus; Ulcer Foot; Ulcer Healing; Diabetic Foot Ulcer; Non-healing Wound; Wound of Skin; Wound; Foot; Tissue Injury
Keywords: Diabetic Ulcer; Diabetic Foot Ulcer; Non-healing Wound; Tissue Engineering; Regenerative Medicine; Decellularized Matrix; Acellular Dermal Matrix; Tissue Allograft; Indigenous Healing; Advanced Wound Care
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer; Diabetic Foot; Foot Injuries | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: An interventional, two-arm, randomized, prospective study of (1) standard of care (control) vs. (2) DermGEN™ - a decellularized dermal matrix (treatment) will be used in the treatment and management of DFU. Patients will be randomized to each arm (n=60 per arm) based on power calculations using data from our Pilot study.
Masking Description: Masking cannot be accomplished as one intervention will require application of an advanced wound care product (DermGEN™) and the other arm (control) will not receive the intervention. This will be quite obvious to all.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): The standard of care includes physical examination, wound debridement, total cast or offloading boot, non-adherent dressing (PolyMem®) for wound covering, weekly visit for ongoing assessment
  Interventions: Procedure: Standard of Care
- DermGEN™ (Experimental): A decellularized dermal matrix created from donated human skin. This arm will receive the same care as the Standard of Care control arm-physical examination, wound debridement, total cast or offloading boot, non-adherent dressing (PolyMem®) for wound covering, weekly visit for ongoing assessment-with the addition of DermGEN™ onto the wound at the first visit.
  Interventions: Other: DermGEN™

INTERVENTIONS:
Procedure: Standard of Care — debridement, wound dressings, offloading
  Arms: Standard of Care
Other: DermGEN™ — Decellularized human dermal matrix created from donated human skin
  Other Names: Acellular Dermal Matrix
  Arms: DermGEN™

SUMMARY:
The study will examine the effectiveness of a decellularized dermal matrix (i.e., DermGEN™) in improving wound healing, quality of life and associated costs of treatment of DFUs in First Nations people living in the Northwestern Ontario Communities. First Nations people with active diabetic foot (DFU) ulcer attending a wound care clinic located at the Rainy River district office. An interventional, two-arm, randomized, prospective study of (1) standard of care (control) vs. (2) DermGEN™ - a decellularized dermal matrix (treatment) will be used in the treatment and management of DFU. Patients will be randomized to each arm (n=60 per arm) based on power calculations using data from our Pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Participant and social support (e.g., family, caregiver) ready and willing to participate and comply with follow-up regime
* Participant willing to be involved in self-care (e.g., keep dressing dry at home) required during treatment
* Participant willing to wear Total Contact Cast (TCC) for wound off-loading during treatment
* Participant or legal representative has read and signed the informed consent form
* Documented stable Type I or II diabetes (HbA1C between 5.0 to 10 mmol/L within 1 month prior to Day 0)
* Ulcer has been present for a minimum of 2 weeks as of Day 0
* Ulcer area is ≥2 cm2 prior to debridement at Day 0 of study
* Ulcer extends through dermis and into subcutaneous tissue but without exposure of muscle, tendon, bone or joint capsule
* Ulcer is free of dead tissue and clinical infection, and is comprised of healthy vascular tissue suitable for skin grafting on Day 0
* Adequate perfusion to the extremity determined by at least one of the following:

Palpable pedal pulses, Transcutaneous oxygen measurement at the dorsum of the foot ≥30 mm Hg, Ankle-brachial index ranging from 0.8 to 1.2, At least biphasic Doppler arterial waveforms at the dorsalis pedis and posterior tibial arteries

Exclusion Criteria:

* The individual has any condition that seriously compromises their capacity to provide consent and answers questions related to this study.
* Untreated infection of soft tissue or bone and/or autoimmune connective tissue disorders
* Ulcer is over Charcot deformity (joints deformity of foot and ankle common in people with diabetes)
* Body mass index ≥50 kg/m2
* Ulcer is not classified as diabetes-related
* Ulcer has tunnels or sinus tracts that cannot be completely debrided
* Medical condition(s) that in the investigators' opinion make the patient inappropriate for study (e.g active liver disease)
* Presence of malignant disease not in remission for 5 years or more
* The individual is undergoing chemotherapy/radiation therapy
* The individual received radiation therapy within 30 days of Day 0 of study
* The individual is taking an immunosuppressant medication (e.g., corticosteroids, immunosuppression or cytotoxic agents), or is anticipated to require such agents during study
* Presence of acute or chronic hepatitis, liver disease, anemia, serum albumin <2.0 gm/dL, or has alkaline phosphatase or LDH at twice the normal upper limit
* Obvious clinical signs and symptoms of ongoing tissue infection (i.e., cellulitis) or bone infection (i.e., osteomyelitis)
* Female individuals are pregnant at time or intend to get pregnant during study time
* The individual has known allergies to antibiotics, such as penicillin and streptomycin
* The individual is an active smoker (smoke one or more cigarette a day)
* The individual has a history of a bleeding disorder or is taking blood thinner medication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean and median reduction in wound area in the first 4 weeks | 4 weeks
  Mean and Median reduction in wound area in comparison to Treatment day 0. Area measured with Silhouette® measurement camera.
Proportion with complete healing in the first 8 weeks | 8 weeks
  Proportion with complete healing in the first 8 weeks. (Complete healing is defined as 100% epithelialization without drainage.)
Proportion with complete healing in the first 12 weeks | 12 weeks
  Proportion with complete healing in the first 12 weeks. (Complete healing is defined as 100% epithelialization without drainage.)
Incidence of adverse events. | Reports included at any time up to and including 20 weeks post treatment.
  Number of adverse events observed for each arm divided by participants in each arm, reported as a percentage
Impact of Treatment on Wound - LUMT Score | 1 week
  Impact of treatment as measured by Leg Ulcer Management Tool (LUMT) score. Comparing initial LUMT score on treatment day 0 to subsequent weeks.
Impact of Treatment on Wound - LUMT Score | 2 weeks
  Impact of treatment as measured by Leg Ulcer Management Tool (LUMT) score. Comparing initial LUMT score on treatment day 0 to subsequent weeks.
Impact of Treatment on Wound - LUMT Score | 3 weeks
  Impact of treatment as measured by Leg Ulcer Management Tool (LUMT) score. Comparing initial LUMT score on treatment day 0 to subsequent weeks.
Impact of Treatment on Wound - LUMT Score | 4 weeks
  Impact of treatment as measured by Leg Ulcer Management Tool (LUMT) score. Comparing initial LUMT score on treatment day 0 to subsequent weeks.
Impact of Treatment on Wound - LUMT Score | 8 weeks
  Impact of treatment as measured by Leg Ulcer Management Tool (LUMT) score. Comparing initial LUMT score on treatment day 0 to subsequent weeks.
Impact of Treatment on Wound - LUMT Score | 12 weeks
  Impact of treatment as measured by Leg Ulcer Management Tool (LUMT) score. Comparing initial LUMT score on treatment day 0 to subsequent weeks.
Impact of Treatment on Wound - LUMT Score | 20 weeks
  Impact of treatment as measured by Leg Ulcer Management Tool (LUMT) score. Comparing initial LUMT score on treatment day 0 to subsequent weeks.
Impact of Treatment on Quality of Life (WoundQoL) | 4 weeks
  Impact of treatment on Quality of Life using the WoundQoL questionnaire score. Comparison of score on treatment day 0 to subsequent weeks.
Impact of Treatment on Quality of Life (WoundQoL) | 8 weeks
  Impact of treatment on Quality of Life using the WoundQoL questionnaire score. Comparison of score on treatment day 0 to subsequent weeks.
Impact of Treatment on Quality of Life (WoundQoL) | 12 weeks
  Impact of treatment on Quality of Life using the WoundQoL questionnaire score. Comparison of score on treatment day 0 to subsequent weeks.
Impact of Treatment on Quality of Life (WoundQoL) | 20 weeks
  Impact of treatment on Quality of Life using the WoundQoL questionnaire score. Comparison of score on treatment day 0 to subsequent weeks.

SECONDARY OUTCOMES:
Proportion with complete healing at any time point | up to and including 20 weeks post initial treatment (Day 0)
  Number of wounds closed (Complete healing is defined as 100% epithelialization without drainage)at any time divided by the number of participants in each arm reported as a percentage
Time to first-measured complete healing | up to and including 20 weeks post initial treatment (Day 0)
  Time to first-measured complete healing (Complete healing is defined as 100% epithelialization without drainage)
Mean and median reduction in wound area at 8 weeks | 8 weeks
  Mean and Median reduction in wound area in comparison to Treatment Day 0. Area measured with Silhouette® measurement camera.
Mean and median reduction in wound area at 12 weeks | 12 weeks
  Mean and Median reduction in wound area in comparison to Treatment Day 0. Area measured with Silhouette® measurement camera.

CONTACTS AND LOCATIONS:
Overall Officials: Paul F Gratzer, Ph.D., Principal Investigator — Dalhousie University
Locations (1):
- Northwestern Ontario (NWO) Wound Care Centre of Excellence, Emo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Site for product description, use — http://decelltechnologies.com